CLINICAL TRIAL: NCT07303946
Title: Double-Blind, Crossover, Feasibility Study of Deep Brain Stimulation of the Anterior Cingulate Bundle (ACB) and the Ventral Anterior Limb of the Internal Capsule (vALIC) in Patients With Intractable Obsessive Compulsive Disorder (OCD)
Brief Title: Deep Brain Stimulation of the Anterior Cingulate Bundle (ACB) and the Ventral Anterior Limb of the Internal Capsule (vALIC) in Patients With Intractable Obsessive Compulsive Disorder (OCD)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Brown University (Other); Baylor College of Medicine (Other); Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5POMH106435P52
Record Dates: First submitted 2022-12-05; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: deep brain stimulation; intractable OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- ACB (Experimental): DBS of the anterior cingulate bundle (ACB)
  Interventions: Device: Medtronic Percept system and 3391 3387 Medtronic DBS electrodes
- vALIC arms (Experimental): DBS of the ventral anterior limb of the internal capsule (vALIC)
  Interventions: Device: Medtronic Percept system and 3391 3387 Medtronic DBS electrodes

INTERVENTIONS:
Device: Medtronic Percept system and 3391 3387 Medtronic DBS electrodes — Surgical implantation of deep brain stimulation electrodes with stimulation at one of two intracranial targets depending on randomization and crossover status.

SUMMARY:
This is a double blind pilot feasibility study, with a within subject crossover design of DBS of the anterior cingulate bundle(ACB) and the ventral anterior limb of the internal capsule(vALIC) in four patients with intractable OCD. Patients will be screened according to inclusion exclusion criteria listed above, approved by an independent Neuropsychiatric review board and informed consent obtained.

DETAILED DESCRIPTION:
This is a double blind pilot feasibility study, with a within subject crossover design of DBS of the anterior cingulate bundle(ACB) and the ventral anterior limb of the internal capsule(vALIC) in four patients with intractable OCD. Patients will be screened according to inclusion exclusion criteria listed above, approved by an independent Neuropsychiatric review board and informed consent obtained. Following implantation of bilateral Medtronic Percept stimulating and recording electrodes in the ACB with electrode Medtronic 3391 and of bilateral Medtronic 3387 electrodes in participants, they will be entered into a two week baseline period with baseline clinical assessments(see Schedule of Assessments) and imaging. Patients will be randomized into ACB or vALIC arms of the study and enter a two week period of stimulation optimization followed by 12 weeks of active blinded treatment in the first condition and then crossed over to the alternate condition where following discontinuation of the first condition stimulation an additional two week period of stimulation optimization in the alternate condition will be followed by an additional twelve weeks of stimulation in the alternate condition. Primary outcome measures will include the YBOCs-II and the Clinical Global Assessment. Ratings will be obtained by independent raters blind to stimulation condition. Following the completion of the second 12 week blinded period, the patient will enter an open nonblinded study of ACB plus vALIC stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. OCD, diagnosed by Structured Clinical Interview for DSM-IV (SCID-IV), judged of disabling severity with a Yale-Brown Obsessive Compulsive Scale (YBOCS) score of at least 30 and a Global Assessment of Functioning (GAF) score of 45 or less.
2. Persistence of severe symptoms and impairment for five or more years despite at least three adequate (≥3 months at the maximum tolerated dose) serotonin transporter inhibitor trials (fluoxetine, sertraline, fluvoxamine, paroxetine, citalopram, escitalopram, or clomipramine) alone or in combination with ii. Adequate behavior therapy (≥20 sessions of expert exposure and response prevention), and iii. Augmentation of one of the selective SRIs with clomipramine, a neuroleptic, and clonazepam.
3. Age between 21 and 65 years.
4. Able to understand and comply with instructions.
5. Able to give fully informed, written consent in the judgment of the site Consent Monitor.
6. Either drug free or on a stable drug regimen for at least 6 weeks.
7. Good general health.
8. A family member or significant other, in contact with the patient every 1-3 days, is available and willing to communicate with the research team if the patient's clinical status worsens, and if necessary to accompany patients to study visits.
9. The local referring psychiatrist is willing to provide ongoing care during and after the trial

Exclusion Criteria:

1. personal/family history (1st/2nd degree relatives) of schizophrenia or schizoaffective disorder, other primary psychotic disorder, bipolar disorder;
2. present PTS;
3. present acute suicidality or suicidal ideation;
4. personal history of head injury, epilepsy, tic or other neurological disorders, neurodevelopmental (e.g., autism), systemic medical (metabolic, endocrine, chronic inflammatory, vascular, autoimmune) disease from medical records and self-report (all of which may confound interpretation of neuroimaging measures);
5. MMSE score < 24;
6. premorbid IQ estimate < 85;
7. visual disturbance (<20/40 Snellen visual acuity, corrected);
8. left/mixed handedness;
9. current, or alcohol or illicit substance abuse/dependence in the last 3 months, determined by clinical assessment and urine toxicology;
10. contraindications to MRI,: metallic foreign objects, e.g., aneurysm clips/pacemakers, or questionable history of metal fragments, claustrophobia raising the risk of panicking in enclosed spaces;
11. positive pregnancy test for women of reproductive age, or women not using medically acceptable birth control throughout the study (barrier and/or oral contraceptives);
12. current psychotic symptoms (potential confounding effect on neuroimaging measures; see above);
13. an increased risk of seizure, determined by history;

4) potentially proconvulsant medications (e.g., bupropion, tricyclic antidepressants, first-generation antipsychotics, lithium), and medications reducing cortical excitability (e.g., anticonvulsants, benzodiazepines, atypical antipsychotics).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) | At the final visit of Stage 1, which occurs at the end of 12 weeks of active stimulation of the first target.
  The Y-BOCS measures obsessive-compulsive symptom severity on a scale of 0-40. Higher scores indicate higher symptom severity (i.e., worse outcomes).
Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) | At the final visit of Stage 2, which occurs at the end of 12 weeks of active stimulation of the second target.
  The Y-BOCS measures obsessive-compulsive symptom severity on a scale of 0-40. Higher scores indicate higher symptom severity (i.e., worse outcomes).
Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) | At the final visit of Stage 3, which occurs at the end of 12 weeks of active stimulation of both targets.
  The Y-BOCS measures obsessive-compulsive symptom severity on a scale of 0-40. Higher scores indicate higher symptom severity (i.e., worse outcomes).
Clinical Global Impression (CGI) | At the final visit of Stage 1, which occurs at the end of 12 weeks of active stimulation of the first target.
  The CGI measures severity of illness and improvement in symptoms since enrollment. Items are each rated on a scale of 1-7. Higher scores indicate worse outcomes.
Clinical Global Impression (CGI) | At the final visit of Stage 2, which occurs at the end of 12 weeks of active stimulation of the second target.
  The CGI measures severity of illness and improvement in symptoms since enrollment. Items are each rated on a scale of 1-7. Higher scores indicate worse outcomes.
Clinical Global Impression (CGI) | At the final visit of Stage 3, which occurs at the end of 12 weeks of active stimulation of both targets.
  The CGI measures severity of illness and improvement in symptoms since enrollment. Items are each rated on a scale of 1-7. Higher scores indicate worse outcomes.

SECONDARY OUTCOMES:
Global Assessment of Functioning (GAF) | At the final visit of Stage 1, which occurs at the end of 12 weeks of active stimulation of the first target.
  The GAF measures overall functioning across multiple life domains. It is rated on a scale of 0-100. Higher scores indicate higher levels of functioning (i.e., better outcomes).
Global Assessment of Functioning (GAF) | At the final visit of Stage 2, which occurs at the end of 12 weeks of active stimulation of the second target.
  The GAF measures overall functioning across multiple life domains. It is rated on a scale of 0-100. Higher scores indicate higher levels of functioning (i.e., better outcomes).
Global Assessment of Functioning (GAF) | At the final visit of Stage 3, which occurs at the end of 12 weeks of active stimulation of the both targets.
  The GAF measures overall functioning across multiple life domains. It is rated on a scale of 0-100. Higher scores indicate higher levels of functioning (i.e., better outcomes).
Sheehan Disability Scale (SDS) | At the final visit of Stage 1, which occurs at the end of 12 weeks of active stimulation of the first target.
  The SDS measures social and occupational functional impairment resulting from psychiatric symptoms. It is rated on a scale of 0-30. Higher scores indicate greater functional impairment (i.e., worse outcomes).
Sheehan Disability Scale (SDS) | At the final visit of Stage 2, which occurs at the end of 12 weeks of active stimulation of the second target.
  The SDS measures social and occupational functional impairment resulting from psychiatric symptoms. It is rated on a scale of 0-30. Higher scores indicate greater functional impairment (i.e., worse outcomes).
Sheehan Disability Scale (SDS) | At the final visit of Stage 3, which occurs at the end of 12 weeks of active stimulation of both targets.
  The SDS measures social and occupational functional impairment resulting from psychiatric symptoms. It is rated on a scale of 0-30. Higher scores indicate greater functional impairment (i.e., worse outcomes).

IPD SHARING:
Plan to Share IPD: No